CLINICAL TRIAL: NCT03826329
Title: Risk Factors of Second Surgery for Adjacent Segment Disease Following Anterior Cervical Discectomy and Fusion: a 16-year Cohort Study
Brief Title: Risk Factors of Second Surgery for Adjacent Segment Disease Following Anterior Cervical Discectomy and Fusion
Acronym: 2nd ACDF
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal Investigator, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2018-09-006CC
Record Dates: First submitted 2019-01-27; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Spinal Fusion
Keywords: Adjacent segment disease (ASD); Second surgery; Anterior cervical discectomy and fusion (ACDF); Risk factors; Cohort study
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: The observational study included all patients who had been admitted for their first ACDF surgery during the 16-year span, began on January 1st, 1998 till the end of 2013, recorded in the NHIRD. The admission for cervical disc herniation and spondylosis were identified using the ICD9-CM diagnostic codes of 722.0, 722.4 and 722.71, while the surgery of ACDF was confirmed with the procedure codes of 80.51, 81.00 and 81.02 during the same hospitalization.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — this is an observational study, there is no intervention in this study

SUMMARY:
Although the incidence of second surgery for adjacent segment disease (ASD) after anterior cervical discectomy and fusion (ACDF) has been reported, its risk factors remain elusive. Few studies have had a sufficiently large number of patients, long follow-up time, and high follow-up rate for investigation. To identify non-surgical risk factors of second surgery for ASD following ACDF, the study used a national cohort with comprehensive follow-up.

DETAILED DESCRIPTION:
All second ACDF surgery after one year from the first ACDF were identified as a consequence of ASD that required another surgery. A multivariate competing risk survival model, Kaplan-Meier survivorship, and average time to events were calculated.

2.1. Data source and ethical concerns The study used the National Health Insurance Research Database (NHIRD), a national database containing 26 million administered insurants accumulated from January 1997 to December 2013, provided by the National Health Research Institutes of Taiwan. Due to the unique social-welfare health insurance system operated by the government, it is mandatory for every resident in Taiwan to be enrolled. Thus, the NHIRD has covered 99% of the population since its launch in 1996. The monopolistic national health insurance also offers unrestricted access to any healthcare provider of the patients' choices. The statistics, therefore, gathered by the NHIRD represent a sound cohort for investigation of the natural course and subsequent management of diseases. It is particularly good for studies that need longitudinal observation for repeat treatment (i.e. surgery for ASD) because it allows for the capture of events, even though they may occur in multiple or different institutes and hospitals. The universal coverage and comprehensive follow-up provided a valuable chance to study ASD.

All the personal information had already undergone a de-identification and encryption process. Individual and hospital identifiers are unique to the research database and researchers therefore cannot trace individual patients or health service providers.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been admitted for their first ACDF surgery during the 16-year span, began on January 1st, 1998 till the end of 2013, recorded in the NHIRD

Exclusion Criteria:

* any re-operation (i.e. ACDF) within 365 days from the indexed date of the first ACDF were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included all patients who had been admitted for their first ACDF surgery during the 16-year span, began on January 1st, 1998 till the end of 2013, recorded in the NHIRD. The admission for cervical disc herniation and spondylosis were identified using the ICD9-CM diagnostic codes of 722.0, 722.4 and 722.71, while the surgery of ACDF was confirmed with the procedure codes of 80.51, 81.00 and 81.02 during the same hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 5565 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
The date of re-operation (Second ACDF) | from patient's index surgery to the end of follow-up (2013/12/31), 4.66 years in average
  Patients were followed-up for the subsequent surgery (second ACDF) after their index operation (first ACDF). We used the hospitalization date of each admission record as the date of outcome (second ACDF). Each patient was followed-up from his index surgery (first ACDF) to re-operation (second ACDF), death, or end of follow-up (2013/12/31) which comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chun Chen, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Yu-Chun Chen, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The PI have no right to share the data